CLINICAL TRIAL: NCT03320642
Title: GRAVITAS-119: A Single-Arm, Open-Label, Phase 1 Study of Itacitinib in Combination With Calcineurin Inhibitor-Based Interventions for the Prophylaxis of Graft-Versus Host Disease
Brief Title: GRAVITAS-119: Itacitinib in Combination With Calcineurin Inhibitor-Based Interventions for the Prophylaxis of Graft-Versus Host Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INCB 39110-119/GRAVITAS-119; 2017-002922-19 (EudraCT Number)
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancies
Keywords: Acute leukemia; chronic myelogenous leukemia; myelodysplasia; chronic lymphocytic leukemia/small lymphocytic lymphoma; follicular; marginal zone; diffuse large B-cell; Hodgkin's lymphoma; mantle cell lymphoma; Janus kinase inhibitor; graft-versus-host disease
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Mantle-Cell; Graft vs Host Disease | interventions — itacitinib; INCB039110; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Itacitinib + Calcineurin Inhibitor (CNI) -Based Interventions (Experimental): Itacitinib in combination with a CNI-based intervention.
  Interventions: Drug: Itacitinib; Drug: Calcineurin inhibitor

INTERVENTIONS:
Drug: Itacitinib — Itacitinib administered orally once daily at the protocol-defined dose.
  Other Names: INCB039110
Drug: Calcineurin inhibitor — The CNI-based prophylaxis regimen will be identified by the investigator before the subject's enrollment and will consist of the combination of tacrolimus/methotrexate, cyclosporine A/mycophenolate mofetil or tacrolimus plus post-treatment cyclophosphamide. Antithymocyte globulin may be included at the treating investigator's discretion with the tacrolimus/methotrexate or cyclosporine A/mycophenolate mofetil combinations.

SUMMARY:
The purpose of this study is to assess the impact and safety of itacitinib in combination with calcineurin inhibitor (CNI)-based interventions for the prophylaxis of graft-versus-host-disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute leukemia, chronic myelogenous leukemia, or myelodysplasia with no circulating blasts and < 5% blasts in the bone marrow.
* Subjects with non-Hodgkin lymphoma, including but not limited to chronic lymphocytic leukemia/small lymphocytic lymphoma, follicular, marginal zone, diffuse large B cell, or mantle cell lymphoma must have chemosensitive disease at time of transplant. Subjects with Hodgkin lymphoma with chemosensitive disease at the time of transplant.
* Must be candidates for reduced-intensity conditioning regimens.
* Must be candidates for peripheral blood stem cell transplants.
* Karnofsky Performance Status score ≥ 70% or Eastern Cooperative Oncology Group Performance Status score of 0 to 2.
* Serum creatinine ≤ 2.0 mg/dL or creatinine clearance ≥ 40 mL/min measured or calculated by Cockcroft-Gault equation.
* Be willing to avoid pregnancy or fathering children.

Exclusion Criteria:

* Has previously received an allogenic hematopoietic stem cell transplant.
* Presence of an active uncontrolled infection.
* Known HIV infection.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment or at risk for HBV reactivation.
* Prior malignancies.
* Severe organ dysfunction.
* Prior treatment with a JAK inhibitor or with an investigational agent, device, or procedure within 21 days of enrollment.
* Currently breastfeeding.
* Known allergies, hypersensitivity, or intolerance to any of the study medications.
* Receipt of live (including attenuated) vaccines during the study, or anticipation of need for such a vaccine during the study.
* History of primary idiopathic myelofibrosis or any severe marrow fibrosis that would prolong neutrophil engraftment to > 28 days after transplant.
* Post-transplant maintenance therapy for the hematologic malignancy or plans to initiate maintenance therapy during study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with hematologic recovery when itacitinib is added to GVHD prophylaxis treatment | Day 28
  Hematologic recovery defined as demonstrating both neutrophil recovery (ANC ≥ 500/mm^3 for 3 consecutive measurements) and platelet recovery (platelet count ≥ 20,000/mm^3 with no requirement for platelet transfusion in the preceding 3 days).

SECONDARY OUTCOMES:
GVHD relapse-free survival rate | Days 100, 180 and 365
  Defined as the proportion of subjects who do not experience Grade III-IV acute GVHD (aGVHD), chronic GVHD (cGVHD) requiring systemic therapy, malignancy relapse or progression, or death due to any cause.
Relapse-free survival | Up to 1 year
  Defined as the interval between enrollment and malignancy relapse or progression, or death, whichever occurs first.
Transplant-related mortality | Up to 1 year
  Defined as the proportion of subjects who die due to causes other than malignancy relapse or progression.
Median time to neutrophil and platelet engraftment | Up to Day 28
  Defined as the median time to achieve neutrophil and platelet engraftment.
Percentage of participants who achieve neutrophil and platelet engraftment | Up to Day 28
  Defined as the median time to achieve engraftment and hematologic recovery at prespecified time points.
Donor Chimerism | Up to Day 28
Proportion of subjects who are diagnosed with Grade II-IV aGVHD, by each grade and by Grade III/IV | Days 100 and Days 180
  Measured to assess the incidence of aGVHD.
Proportion of subjects who are diagnosed with cGVHD by grade (mild, moderate, or severe) | Up to 1 year
  Measured to assess the incidence of cGVHD.
Infection rate | Up to 1 year
  Defined as the proportion of subjects who demonstrate an infection and/or cytomegalovirus reactivation.
Overall survival | Up to 1 year
  Defined as the interval between enrollment and death due to any cause.
Participants with Grade 3-5 treatment-emergent adverse events (TEAEs) | Up to approximately 200 days
  TEAE is defined as either an adverse event (AE) reported for the first time or worsening of a pre-existing condition after the first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, MD, Study Director — Incyte Corporation
Locations (17):
- United States (9):
  - Anschutz Cancer Pavilion - University of Colorado, Aurora, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - Chru de Lille Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Chu Vandoeuvre-Les-Nancy, Hopital Brabois, Vandœuvre-lès-Nancy
- Italy (3):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni Xxiii (Presidio Papa Giovanni Xxiii), Bergamo
  - Azienda Ospedaliera San Gerardo Di Monza, Monza
  - Comitato Di Bioetica Della Fondazione Irccs Policlinico San Matteo, Pavia
- Spain (2):
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No